CLINICAL TRIAL: NCT00053222
Title: A Phase II Study Of Arsenic Trioxide In Patients With Adenocarcinoma Of The Pancreas Refractory To Gemcitabine
Brief Title: Arsenic Trioxide in Treating Patients With Pancreatic Cancer That Has Not Responded to Gemcitabine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11839A; UCCRC-11839A; NCI-5839
Record Dates: First submitted 2003-01-27; First posted 2003-01-28 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Pancreatic Cancer
Keywords: recurrent pancreatic cancer; stage II pancreatic cancer; stage III pancreatic cancer; adenocarcinoma of the pancreas; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Arsenic Trioxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm A (Experimental): Arsenic trioxide (0.3 mg/kg/day iv for 5 days every 28 days)
  Interventions: Drug: arsenic trioxide

INTERVENTIONS:
Drug: arsenic trioxide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of arsenic trioxide in treating patients who have locally advanced or metastatic pancreatic cancer that has not responded to gemcitabine.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the objective response rate to arsenic trioxide in patients with pancreatic cancer who have progressed after first-line treatment with a gemcitabine-containing regimen when treated with arsenic trioxide.
* Determine the toxicity of this drug in these patients.
* Determine the duration of response, median and overall survival, and time to progression in patients treated with this drug.

OUTLINE: This is a multicenter study.

Patients receive arsenic trioxide IV over 1 hour on days 1-5. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients are followed for survival.

PROJECTED ACCRUAL: A total of 12-37 patients will be accrued for this study within 9-12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed adenocarcinoma of the pancreas

  * Locally advanced or metastatic disease
* Unidimensionally measurable disease

  * At least 1 lesion that is at least 20 mm with conventional techniques or at least 10 mm with spiral CT scan
* Must have progressed after chemotherapy with a gemcitabine-containing regimen
* No known brain metastases

PATIENT CHARACTERISTICS:

Age

* Over 18

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin no greater than 1.5 mg/dL
* AST/ALT no greater than 5 times upper limit of normal

Renal

* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance at least 60 mL/min

Cardiovascular

* QTc less than 500 msec at baseline by EKG
* No New York Heart Association class III or IV heart failure
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior allergic reactions attributed to compounds of similar chemical or biological composition to arsenic trioxide
* No other active malignancy within the past 5 years except nonmelanoma skin cancer or carcinoma in situ of the cervix
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance
* No other uncontrolled illness

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent immunotherapy
* No concurrent colony-stimulating factors during the first course of the study

Chemotherapy

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* No prior arsenic trioxide
* No other concurrent chemotherapy
* No more than 1 prior chemotherapy regimen for metastatic disease

Endocrine therapy

* No concurrent hormonal therapy

Radiotherapy

* At least 4 weeks since prior radiotherapy and recovered
* No concurrent therapeutic radiotherapy

Surgery

* At least 4 weeks since major surgery

Other

* No other concurrent investigational or commercial anticancer agents or therapies
* No other concurrent investigational agents
* No concurrent antiretroviral therapy in HIV-positive patients
* No concurrent medications for other comorbid conditions that are known to prolong the QT interval

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2003-02; Primary Completion 2005-01 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Objective response | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Hedy L. Kindler, MD, Study Chair — University of Chicago
Locations (11):
- United States (11):
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Evanston Northwestern Health Care - Evanston Hospital, Evanston, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - LaGrange Memorial Hospital, LaGrange, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Oncology/Hematology Associates of Central Illinois, P.C., Peoria, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Fort Wayne Medical Oncology and Hematology, Incorporated, Fort Wayne, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Lakeland Cancer Care Center at Lakeland Hospital - St. Joseph, Saint Joseph, Michigan